CLINICAL TRIAL: NCT07290088
Title: An Open Label, Multicenter, Safety and Efficacy Phase II/III Study of PRL3-Zumab in Solid Tumor Patients
Brief Title: Phase II/III Trial of PRL3-Zumab in Advanced Solid Tumor Patients
Acronym: PRL3-zumab
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Intra-IMMUSG Pte Ltd (Industry)
Collaborators: Kuala Lumpur General Hospital (Other Government); Beacon Hospital (Other); Hospital Universiti Sains Malaysia (Other); University Malaysia Medical Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 226688-M
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: PRL3-ZUMAB Monotherapy (Other): Single Arm
  Interventions: Biological: PRL3-ZUMAB

INTERVENTIONS:
Biological: PRL3-ZUMAB — PRL3-zumab will be administered every 2-week/dose till patient progress or develops intolerable toxicity or withdraw consent.
  A dose at 10-days is allowed at the first 4 doses when patients had heavier tumor burden since PRL3-zumab PK t ½ = 12 days (±2 days).

SUMMARY:
This is a Multi-Center, Phase II/III, open-label, single dose level (6 mg/kg) basket trial of PRL3-zumab monotherapy in solid cancer patients.

The study will consist of a Screening Period (Day - 14 to Day -1) for completion of all screening assessments before the first administration of study treatment, a Treatment Period during which visits will occur every 2-week (PK T1/2 = 12 days ±2 days), once the decision to discontinue treatment for any reason, an End of Treatment (EOT) visit will be performed within 14 days ±4 days after last dose of study treatment. Safety Follow-up/EOS visit will be performed 28 days ±2 days after last dose of study treatment and survival follow-up call will be performed every month up to 6 months after EOS visit.

PRL3-zumab will be administered by intravenous (i.v.) infusion till patient meets discontinuation criteria (progressive disease, clinically or per iRECIST, intolerable toxicity or withdrawal of consent). One cycle of treatment will be 4-weeks (2 infusions, 12 days±2 days apart). Patients will undergo safety assessment including laboratory tests prior to each infusion. Efficacy will be assessed by iRECIST at baseline and every 4 doses after study treatment. QoL assessments will be performed at Screening and every 4 doses ±7 days during treatment. A patient will be discontinued from study treatment if the patient progress clinically or per iRECIST criteria, or for intolerable toxicity, or if the patient withdraws consent. An EOT visit will be performed within14 days ±4 days after last study treatment dose.

DETAILED DESCRIPTION:
Safety:

Patient safety will be evaluated based on physical examination, vital signs (blood pressure [systolic and diastolic], heart rate, respiratory rate, and temperature), clinical laboratory tests (hematology, clinical chemistry, coagulation) and adverse events per CTCAE v5. Patient safety will be assessed on an ongoing basis during each cycle.

Quality of life assessment EQ-5D and EORTC-QLQ-C30 questionnaire scores will be obtained at Screening and every 2 cycles (8 weeks ± 2 days) for C1 to C4 and 8 weeks ±7 days for the rest of the scheduled visits) for the duration of the study.

DURATION OF THE STUDY:

The planned duration of the treatment is till patient meets discontinuation criteria. In addition, the study includes a patient enrolment period of 14 days, EOT visit within 14 days after last dose of study treatment and an EOS visit for safety follow-up 28 days after the last dose of study treatment. Survival study follow-up call will be done monthly till 6 months after EOS visit.

Cycle Period Per Treatment:

One cycle of treatment will be 2 infusions administration (4-week) (PK T1/2= 12 days ±2 days for each infusion).

Treatment Period:

PRL3-zumab will be administered till progression of disease (iRECIST or clinical criteria), intolerable toxicity or withdrawal of consent.

STATISTICAL CONSIDERATIONS:

Sample Size Determination Sample size: for alpha, α = 0.05 and power, β = 0.9 PRL3-zumab therapy: 30% PRL3-zumab therapy min response rate: 10% Number of patients in each arms (treatment group) for phase II (Stage): 22 Response R: 2 No patients in each arms (treatment group): 33 Response R: 6 Total patients adjusted for 10% dropout:42 Total patients adjusted for 20% dropout: 52

Sample size was estimated based on the primary efficacy parameter, which is the PFS or TTP as per iRECIST criteria base on the investigator's assessment of tumor response for patients with PRL3-zumab. The tumor response of the Solid Tumor is defined as Progression Free Survival (PFS) or Time to progression (TTP) with minimum survival of 6 months.

Assume an overall response rate of 30% to PRL3-zumab therapy and there will be no further interest in this combination treatment if the response rate was as low as 10% (less than half the treated patients).

By using the Simon's minimax design with type 1 and type 2 errors of 0.05 and 0.1, 22 patients will be enrolled in stage 1 (Phase 2), requiring at least 2 responses before proceeding to enroll an additional 11 patients in stage 2 (Phase 3).

Therefore, a total of 33 patients will be enrolled. PRL3-zumab will be rejected as ineffective if less than 6 out of the total of 33 patients responded to PRL3-zumab therapy.

Taking into account of drop-out rate of 10%, total of 42 patients will be enrolled.

Taking into account of drop-out rate of 20%, total of 52 patients will be enrolled.

Primary endpoint is solid tumor response to PRL3-zumab. Solid tumor respond is define as patients who has achieve Progression Free Survival (PFS) or Time to Progression with minimum 6 months. Progression Free Survival is defined as the time from random assignment to disease progression or death in any cause.

PRL3-zumab is a novel unconventional cancer immunotherapy behind Standard of Care (SOC), we will follow the protocol to recruit ~ 33 patients with life expectancy > 6-month survival for 12 doses to be evaluated at three time points: > 4, > 8, >12 doses respectively for PFS/TTP.). Patients who do not have at least one evaluable post-baseline tumor assessment (< 4 doses) will be replaced .

Clinical benefits related to tumor sizes, blood tests, cancer markers will be analyzed back to back within the same patients.

The objectives are to identify patients who will respond to PRL3-zumab better than their own prior lines of SOCs. Since PRL3-zumab is a single arm/monotherapy trial, we will also compare with historical data as additional control arms of drug efficacy study.

An interim analysis will be conducted for efficacy and safety when approximately 30 patients completed the minimum 6 months follow-up with 22 evaluable patients. The result of the phase II analysis requiring at least 2 responses before proceeding to enroll an additional 11 patients to proceed with phase III.

Efficacy Analyses:

The primary efficacy endpoint is the PFS or TTP as per iRECIST criteria based on the Investigator's assessment of tumor response. The count and percentage of patients with responses along with the corresponding 95% confidence interval will be calculated and presented.

Secondary efficacy endpoints will be analyzed as follows:

CBR will be analyzed using the same methodology as for the primary efficacy endpoint.

Counts and percentages of patients with responses, along with exact 95% CI will be presented. CBR is defined as the percentage of patients who have achieved CR, PR, or SD at > 4 doses, 8 doses, and 12 doses during the Treatment Period as per iRECIST criteria based on Investigator's assessment.

Safety Analysis:

AEs will be classified according to CTCAE v5 or the latest version. Treatment-emergent adverse events (TEAEs), Treatment-related TRAEs, serious TEAEs, TEAE of Grade 2 or greater, TEAEs leading to death, TEAEs leading to treatment discontinuation, and TEAEs leading to dose modification will be summarized respectively. Clinical laboratory data, vital signs, and ECOG PS will be summarized descriptively. Physical examinations findings will be presented in a listing.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 - 75 years with solid tumors
2. Willing to provide written informed consent for the study.
3. Histopathological diagnosis and metastatic status cancer at study entry.
4. Stage 1-3 patients with no more than 3 prior lines of treatment
5. Life expectancy of more than 6 months (especially for Pancreatic cancer patients).
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
7. Patient should have recovered from toxicity of prior treatment regimen to Grade 1 level except for alopecia or peripheral neuropathy or fatigue as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.
8. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at study entry and must follow highly effective contraception
9. Adequate organ and hematological function as evidenced by the following laboratory studies within 10 days of treatment:

   * Absolute neutrophil count ≥ 1.0 x 109/L.
   * Platelet count ≥ 75 x 109/L. Hemoglobin ≥ 90 g/L (9 g/dL).
   * Prothrombin time and activated partial thromboplastin time ≤ 1.5 x upper limit of normal (ULN) per institutional laboratory normal range.
   * Total bilirubin ≤ 1.5x ULN.
   * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal (ULN) (≤ 5 x ULN in the presence of liver metastases).
   * For patients with hepatocellular carcinoma (HCC) Child Pugh score of ≤ B7.
   * Creatinine < 1.5x ULN.
10. Measurable disease by iRECIST.
11. No history of active hepatitis B or C infection.

Exclusion Criteria:

1. Patient has known untreated or symptomatic central nervous system metastasis.
2. Female patient is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and for 150 days (for pregnancy or conception) or 30 days (for breastfeeding) after the last dose of study treatment.
3. Patient has known history of human immunodeficiency virus (HIV) infection (HIV-1 or HIV-2 antibodies).
4. Patient is receiving systemic glucocorticoids (only if higher than 10 mg or equivalent of prednisolone daily) or other immunosuppressive treatment for autoimmune disease or any other medical condition.
5. Patient has experienced a severe hypersensitivity reaction to another monoclonal antibody.
6. Patient has received treatment with any systemic anti-cancer therapies within 3 weeks prior to starting study treatment.
7. Patient has undergone radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study treatment.
8. Patient is unable to provide informed consent.
9. Patient has received a prior stem cell or bone marrow transplant.
10. Patient with abnormal cachexia.
11. Patient with distended abdomen from ascites.
12. Patient is currently participating in a treatment study or has participated in a study of an investigational agent within 4 weeks prior to the anticipated first dose of study treatment in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Time Frame: From the date of first dose of study drug until first documented disease progression or date of death from any cause, whichever comes first, assessed up to 12 months.
  PFS is defined as the time from the initiation of study treatment to the date of disease progression as per RECIST v1.1 and iRECIST criteria.
Time to Progression (TTP) | From the date of first dose of study drug until first documented disease progression, assessed up to 12 months.
  TTP is defined as the time from the the initiation of study treatment to the date of disease progression as per RECIST v1.1 and iRECIST criteria which does not include deaths.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | Time Frame: From date of first dose of study drug until first documented disease progression or date of death, whichever comes first, assessed at every 8 weeks up to 48 weeks.
  CBR is defined as the percentage of patients with CR, PR, or stable disease (SD) as per RECIST v1.1 and iRECIST criteria based on Investigator's assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Qi Zeng, Study Director — Intra-IMMUSG Pte Ltd
Locations (4):
- Malaysia (4):
  - Hosp. Universiti Sains Malaysia (HUSM), Kelantan, Kota Bharu
  - Beacon Hospital, Kuala Lumpur
  - Hosp. Kuala Lumpur, Kuala Lumpur
  - University Malaysia Medical Centre, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park DJ, Thura M, Chiu VK, Vicuna B, Ang KH, Sanchez B, Chia PL, Kuan KY, Li J, Zhang K, Zheng WH, Hsien Ng MC, Zeng Q. The PRL3-zumab paradigm: A multicenter, single-dose-level phase 2 basket clinical trial design of an unconventional cancer immunotherapy. Cell Rep Med. 2025 May 20;6(5):102120. doi: 10.1016/j.xcrm.2025.102120. Epub 2025 May 8. PMID 40345181
- [Background] Loh AHP, Thura M, Gupta A, Tan SH, Kuan KKY, Ang KH, Merchant K, Chang KTE, Yon HY, Chen Y, Cheng MHW, Mahadev A, Ng MCH, Seng MS, Iyer P, Chia PL, Soh SY, Zeng Q. Exploiting frequent and specific expression of PRL3 in pediatric solid tumors for first-in-child use of PRL3-zumab humanized antibody. Mol Ther Oncolytics. 2023 Aug 18;30:153-166. doi: 10.1016/j.omto.2023.08.006. eCollection 2023 Sep 21. PMID 37674627
- [Background] Chee CE, Ooi M, Lee SC, Sundar R, Heong V, Yong WP, Ng CH, Wong A, Lim JSJ, Tan DSP, Soo R, Tan JTC, Yang S, Thura M, Al-Aidaroos AQ, Chng WJ, Zeng Q, Goh BC. A Phase I, First-in-Human Study of PRL3-zumab in Advanced, Refractory Solid Tumors and Hematological Malignancies. Target Oncol. 2023 May;18(3):391-402. doi: 10.1007/s11523-023-00962-w. Epub 2023 Apr 15. PMID 37060431
- [Background] Thura M, Ye Z, Al-Aidaroos AQ, Xiong Q, Ong JY, Gupta A, Li J, Guo K, Ang KH, Zeng Q. PRL3 induces polypoid giant cancer cells eliminated by PRL3-zumab to reduce tumor relapse. Commun Biol. 2021 Jul 29;4(1):923. doi: 10.1038/s42003-021-02449-8. PMID 34326464
- [Background] Thura M, Al-Aidaroos AQ, Gupta A, Chee CE, Lee SC, Hui KM, Li J, Guan YK, Yong WP, So J, Chng WJ, Ng CH, Zhou J, Wang LZ, Yuen JSP, Ho HSS, Yi SM, Chiong E, Choo SP, Ngeow J, Ng MCH, Chua C, Yeo ESA, Tan IBH, Sng JXE, Tan NYZ, Thiery JP, Goh BC, Zeng Q. PRL3-zumab as an immunotherapy to inhibit tumors expressing PRL3 oncoprotein. Nat Commun. 2019 Jun 6;10(1):2484. doi: 10.1038/s41467-019-10127-x. PMID 31171773
- [Background] Thura M, Al-Aidaroos AQO, Yong WP, Kono K, Gupta A, Lin YB, Mimura K, Thiery JP, Goh BC, Tan P, Soo R, Hong CW, Wang L, Lin SJ, Chen E, Rha SY, Chung HC, Li J, Nandi S, Yuen HF, Zhang SD, Guan YK, So J, Zeng Q. PRL3-zumab, a first-in-class humanized antibody for cancer therapy. JCI Insight. 2016 Jun 16;1(9):e87607. doi: 10.1172/jci.insight.87607. PMID 27699276
- [Background] Guo K, Li J, Tang JP, Tan CP, Hong CW, Al-Aidaroos AQ, Varghese L, Huang C, Zeng Q. Targeting intracellular oncoproteins with antibody therapy or vaccination. Sci Transl Med. 2011 Sep 7;3(99):99ra85. doi: 10.1126/scitranslmed.3002296. PMID 21900592